CLINICAL TRIAL: NCT03087877
Title: Evaluation of the Dexcom G6 Continuous Glucose Monitoring System With a Non-Interferent Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL902020
Record Dates: First submitted 2017-02-24; First posted 2017-03-23 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: The system will be blinded to the user, i.e. no glucose values will be displayed to the subject during the study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CGM Users (Other): Prospective, non-randomized, single-arm. Continuous Glucose Monitoring. Acetaminophen challenge is the intervention.
  Interventions: Device: Acetaminophen Challenge (G6 CGM)

INTERVENTIONS:
Device: Acetaminophen Challenge (G6 CGM) — Evaluation of acetaminophen effect on CGM glucose sensing

SUMMARY:
The objective of the study is to demonstrate effectiveness of the G6 sensor membrane, in preventing acetaminophen's interference effect on glucose sensing.

DETAILED DESCRIPTION:
The interference effect of the sensor will be evaluated by comparing the bias in the glucose values exhibited from the G6 CGM system after administration of acetaminophen. Bias will be evaluated by comparing CGM values to a laboratory referenceusing venous sample measurements.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Diagnosis of diabetes

Exclusion Criteria:

* Pregnancy
* Known gastroparesis
* Abnormal liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-03-04 (Actual); Study Completion 2017-03-04 (Actual)

PRIMARY OUTCOMES:
Interference Effect for the G6 CGM | 6 hrs post dose
  Bias of sensor to reference measurement pre and post acetaminophen administration

SECONDARY OUTCOMES:
Mean of sensor minus YSI values (bias) for various time periods | 6 hrs post dose
  Bias calculated for pre-dose, post dose and peak post dose
Duration of interference effect for the G6 CGM | 6 hrs post dose
  Length of time the inhibition effect is more than 10 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Director — DexCom, Inc.
Locations (4):
- United States (4):
  - AMCR, Escondido, California
  - William Sansum Diabetes Center, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Rainier Clinical Research Center Inc, Renton, Washington

IPD SHARING:
Plan to Share IPD: No